CLINICAL TRIAL: NCT06868121
Title: Assessing the Impact of a Web-based Educational Program on the Sexual Health Outcomes of Young Adult Female Cancer Survivors ~ A Pilot Trial
Brief Title: AYA OMGYES Sexual Health Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB24-0909
Record Dates: First submitted 2025-02-26; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Sexual Dysfunction
MeSH Terms: conditions — Sexual Dysfunction, Physiological

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Delayed Intervention (Other): The delayed intervention group will initially undergo 5 weeks of active observation prior to intervention administration.
  Interventions: Other: OMGYES.com
- Immediate Intervention (Experimental): The immediate intervention group will be administered the intervention at study enrollment.
  Interventions: Other: OMGYES.com

INTERVENTIONS:
Other: OMGYES.com — OMGYES.com is an interactive website that offers information, video tutorials, interviews, tips, and resources to explore female sexual pleasure through groundbreaking research that's told through the real-life experiences of women of all ages and life stages.

SUMMARY:
The purpose of this study is to assess the impact of the web-based intervention OMGYES.com on sexual dysfunction in young adult (YA) female-bodied cancer survivors. This pilot trial seeks to evaluate the intervention's:

* feasibility
* acceptability
* appropriateness.

Researchers will utilize an active observation period to compare outcomes between those receiving the intervention immediately and those who haven't

Participants will:

* Complete online modules at home
* Visit the clinic every 5 weeks for questionnaires

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 40 years
* Diagnosis of cancer between the ages of 15 and 40
* Female genitalia, regardless of gender
* Diagnosed with sexual dysfunction
* Complete Remission and at least two months from a major treatment
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Ability to participate in study modules and to respond to surveys
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients receiving other investigational agents
* Patients expected to be neutropenic or have a significantly high infection risk that would exclude them from vaginal penetration
* Patients who are unable complete the study intervention or surveys

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-16 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of OMGYES.com using the Feasibility of Intervention Measure (FIM) | End of Study (Week 6)
  The Feasibility of Intervention Measure (FIM) is a validated questionnaire that utilizes a 5-point Likert scale to evaluate the extent at which an intervention can be successfully used in a clinical setting.

SECONDARY OUTCOMES:
Acceptability of OMGYES.com using the Acceptability of Intervention Measure (AIM) | End of Study (Week 6)
  The Acceptability of Intervention Measure (AIM) is a validated questionnaire that utilizes a 5-point Likert scale to evaluate the extent to which participants deem an intervention agreeable, palatable, or satisfactory.
Appropriateness of OMGYES.com using the Appropriateness of Intervention Measure | End of Study (Week 6)
  The Acceptability of Intervention Measure (AIM) is a validated questionnaire that utilizes a 5-point Likert scale to evaluate the perceived fit, relevance, or compatibility of an intervention for a given population; and/or perceived fit of the intervention to address a particular issue or problem

CONTACTS AND LOCATIONS:
Overall Officials: Adam DuVall, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Hospital, Chicago, Illinois, United States